CLINICAL TRIAL: NCT02233829
Title: Dopamine Rhythms in Health and Addiction
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No enrollment, delay with drug availability.
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 140187; 14-AA-0187
Record Dates: First submitted 2014-09-06; First posted 2014-09-09 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cocaine Abuse
Keywords: C-11 Raclopride; PET; Circadian Rhythm
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Evening MRI/PET/Raclopride/IV Methylphenidate Session (Active Comparator): The PET [11C] raclopride scan will be done between 5-7 PM. After iv catheters are inserted blood sampling starts and continues throughout study. Cardiac monitoring is initiated and continues until physician discontinues post PET scan. Bolus-plus-infusion method for [11C]raclopride and the administration of intravenous MP (0.5 mg/kg) forty-five minutes after initial bolus injection of [11C]raclopride. Scan to be done for a total of 100 minutes.
  Interventions: Drug: Brain Dopamine Reactivity; Radiation: Brain Dopamine Receptor
- Morning MRI/PET/Raclopride/IV Methylphenidate Session (Active Comparator): Morning Session [11C]raclopride PET scan: To be started between 7-8 AM. After iv catheters are inserted, genetic blood samples are drawn and then blood sampling starts and continues throughout study. Cardiac monitoring is initiated and continues until physician discontinues post PET scan. Bolus-plusinfusion method for [11C]raclopride and the administration of intravenous MP (0.25 mg/kg) fortyfive minutes after initial bolus injection of [11C]raclopride. Scan to be done for a total of 100 minutes.
  Interventions: Drug: Brain Dopamine Reactivity; Radiation: Brain Dopamine Receptor

INTERVENTIONS:
Drug: Brain Dopamine Reactivity — IV methylphenidate, used under IND #124, 912 is injected into the subject s bloodstream to be used in conjunction with PET imaging to show displacement of [11C]raclopride.
Radiation: Brain Dopamine Receptor — The radiotracer [11C] raclopride is used for imaging dopamine receptors and dopamine release.

SUMMARY:
Background:

- Dopamine is a chemical signal linked to the rewarding effects of drugs. Certain genes make these effects sensitive to the time of day they are taken. Cocaine can affect these genes in the brain. Researchers want to measure brain dopamine at different times of day.

Objectives:

- To look for changes to a person s biological clock in the function of the dopamine reward system. To test if cocaine disrupts this.

Eligibility:

* Adults age 21-55 with a cocaine use disorder.
* Healthy volunteers age 21-55.

Design:

* Participants will be screened with medical history, physical exam, interview, and blood and urine tests. Their breath will be tested for alcohol and recent smoking.
* Participants will have 3 overnight clinic visits.
* Visit 1: They will have blood and urine collected and a heart test.
* A plastic tube (catheter) will be placed into a vein in each arm by needle.
* Participants will have a PET scan in a donut-shaped machine. They will lie on a bed that slides in and out of it, wearing a cap. A radiotracer (measures dopamine) and a drug (blocks dopamine removal) will be injected via catheter. Vital signs will be measured and blood will be drawn throughout.
* Visit 2: repeats Visit 1, except at night.
* Visit 3, participants will have urine collected.
* They will have MRI scans in a metal cylinder surrounded by a magnetic field. They will lie on a table that slides in and out of it, with a coil over their head.
* Participants may answer questions, take computer or paper tests, and perform simple actions.
* For 1 week, participants will wear a wrist device that measures daily activity.

DETAILED DESCRIPTION:
Objectives:

The primary objective is to assess if there is disruption of circadian DA rhythms in cocaine addiction. The secondary objective is to assess if dopamine modulates the sensitivity of the brain reward network in a circadian dependent manner.

Study Population:

Non-treatment seeking cocaine abusers (moderate or severe cocaine use disorder as per DSM-IV or DSM 5) and healthy controls. Males and females will be included.

Design:

Participants will undergo two PET scans with [11C]raclopride using a bolus infusion paradigm to assess baseline D2R availability followed by an infusion to assess changes in DA as measured by [11C]raclopride s displacement following an intravenous injection of methylphenidate (MP). They will also undergo a total of 4 MRI scans, two after placebo and two after MP to assess the circadian variations in the sensitivity of the brain reward network. The two [11C]raclopride scans will be done on separate days at least one week apart, one in the morning starting between (7-9 AM) and one in the early evening (5-7 PM) and they will be followed by an MRI scan to assess the sensitivity of the brain reward network under the influence of MP in the morning (9-11AM) and in the evening (7-9 PM). For the Placebo MRI scans participants will be tested either on separate days or on the morning of the evening session or on the evening prior to the morning session. We will use the MRI scans to assess the sensitivity of the brain reward circuit to visual presentation of drug or food cues and to evaluate resting functional connectivity.

Outcome Parameters:

Main outcome measure is to assess if there are differences in DA release between the morning and the evening (displacement of [11C]raclopride binding after MP) and to determine if these diurnal patterns differ in cocaine addiction. Secondary outcome measures are: To assess if DA signaling correlates with reactivity of brain regions to exposure of food and drug cues and with functional connectivity of the reward network and to assess if the reactivity of the reward network shows circadian variability. We will also assess if differences in DA signaling between morning and evening correlate with circadian typology and with measures of spontaneous motor activity and with sleeping patterns.

ELIGIBILITY:
* INCLUSION CRITERIA - ALL PARTICIPANTS:

  1. Between 21 and 55 years of age.
  2. Ability to provide written informed consent.

INCLUSION CRITERIA - SPECIFIC FOR COCAINE USE DISORDER (CUD) PARTICIPANTS:

1. DSM-IV or DSM-5 diagnosis of a moderate or severe cocaine use disorder established through history and clinical exam.
2. Non-treatment seeking cocaine users (actively consuming cocaine - last use within one week of study as assessed by self-reports).
3. Minimum 10 years history of cocaine abuse predominantly via smoking or injection - self-report.
4. Must consume at least 4 grams of cocaine per week - self-report.

EXCLUSION CRITERIA - ALL PARTICIPANTS:

1. Unwilling or unable to refrain from use within 24 hours of scheduled study procedures: psychoactive medications or medications that may affect study results e.g., antibiotics (must finish course at least 24 hours prior to a scheduled procedure), antidiarrheal preparations, anti-inflammatory drugs [systemic corticosteroids are exclusionary], anti-nausea, cough/cold preparations) (self-report, medical history). The following medications are allowable for entry on this study: analgesics (non-narcotic and narcotic for OUD participants); antacids; antiasthma agents that are not systemic corticosteroids; antifungal agents for topical use; antihistamines (non-sedating); H2-Blockers/PPI (proton pump inhibitors); laxatives. The use of antihyperlipidemics and/or diuretics are permitted if they have been taken for at least 1 month before procedure visits and dose has been stabilized as determined by medical history and physical exam. The episodic use of benzodiazepines such as alprazolam ((TM)Xanax), diazepam ((TM)Valium) and lorazepam ((TM)Ativan), will not exclude participants from this study unless they have been taken within the last 24 hours prior to the study.
2. Current or past DSM-IV or DSM-5 diagnosis of a psychiatric disorder (other than cocaine for the cocaine abusers, and nicotine/caffeine for any of the participants) that required hospitalization (any length), or chronic medication management (more than 4 weeks) and that could impact brain function at the time of the study as determined by history and clinical exam.
3. The following current chronically used medications are exclusionary from the study: stimulant or stimulant-like medications (amphetamine, methylphenidate, modafinil) ; analgesics containing narcotics (for controls only); anorexics (sibuteramine); antianginal agents; antiarrhythmics; antiasthma agents that are systemic corticosteroids; antibiotics; anticholinergics; anticoagulants; anticonvulsants; antidepressants; antidiarrheal preparations; antifungal agents (systemic); antihistamines (sedating); antihypertensives; anti-inflammatory drugs (systemic); antineoplastics; antiobesity; antipsychotics; antivirals (except for treatment of HSV with agents without CNS activity, e.g. acyclovir, ganciclovir, famciclovir, valacyclovir); anxiolytics (benzodiazepine or barbiturates); hormones (exceptions: thyroid hormone replacement, oral contraceptives, and estrogen replacement therapy); insulin; lithium; muscle relaxants; psychotropic drugs not otherwise specified (nos) including herbal products (no drugs with psychomotor effects or with anxiolytics, stimulant, antipsychotic, or sedative properties); sedatives/hypnotics. Note that nicotine and/or caffeine use will not exclude participants and that the use of cocaine will not exclude participants with CUD.
4. Major medical problems that can permanently impact brain function (e.g., CNS including seizures and psychosis; cardiovascular including hypertension [BP > 140/90] and clinically significant arrhythmias except bradycardia; metabolic, autoimmune, endocrine; +HIV) as determined by history.
5. Any clinically significant laboratory finding as determined during the screening procedures that could impact brain function or study procedures as evidenced from clinical laboratory results. Since half of the participants in the study will have a diagnosis of cocaine use disorder (CUD), we expect some clinically significant findings that would reflect their recent cocaine use. As an example, a participant might have a mildly elevated Creatinine Kinase as a result of recent cocaine use. The test would reflect an acute rhabdomyolysis due to recent cocaine use, and it would be clinically significant. Nevertheless, if it is a mild episode as expected with cocaine use, it would not affect brain functioning or increase the risk of the procedures for the participants in the study. Therefore, not all abnormal laboratory findings that have clinical significance will be excluded. If a finding reflects altered brain function (e.g., arrhythmias or renal failure) it will be exclusionary for the study.
6. Have had previous radiation exposure (from X-rays, PET scans, or other exposure) that, with the exposure from this study, would exceed NIH annual research limits as determined by medical history and physical exam.
7. Head trauma with loss of consciousness for more than 30 minutes as determined by medical history and physical exam.
8. Pregnant or breast feeding: Females must have negative urine pregnancy test and are not currently breastfeeding. Post-menopausal or surgically sterile (tubal ligation or hysterectomy); or not sexually active with a male partner and able to get pregnant; or documented agreement to use an effective form of birth control. Acceptable forms of contraception include: hormonal contraceptives (birth-control pills, injectable hormones, vaginal-ring hormones); IUD; diaphragm with spermicide; condom with spermicide.
9. History of coagulation disorder as evidenced from clinical laboratory results, medical history.
10. History of glaucoma as determined by medical history. Since glaucoma is screened for clinically at about the age of 40, any subjects 40 or older will undergo a glaucoma screening test if they have not been tested by their primary care physician. A result of 21 mmHg or higher will exclude.
11. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces - self-report checklist.
12. Personal or family history for cerebral aneurism.
13. Past or present history of chest pain and trouble breathing with activity.
14. Diabetes as assessed by medical history.
15. High risk for silent heart diseases as evidenced by high levels of high-sensitivity C-reactive protein or homocysteine in blood, or being overweight or obese. In addition patients with high cholesterol or a family history of heart disease will be evaluated by a cardiologist to determine their eligibility for participation. The cardiologist might request additional tests if he deems it necessary to ensure fitness for participation (ie treadmill stress test). Specifically the cardiologist involved will review the findings of 1) an inability to reach these endpoints, 2) the development of chest pain, 3) significant ST segment changes, 4) significant arrhythmias, and 5) an inability to appropriately increase blood pressure or heart rate with exercise in order to determine if the participant is suitable for inclusion in the study.
16. Cannot lie comfortably flat on your back for up to 2 hours in the PET and MRI scanners - self-report.
17. Weight > 400 pounds which is the maximum weight the PET scanner can hold.
18. Study investigators and staff, as well as their superiors, subordinates and immediate family members (adult children, spouses, parents, siblings).

    * Note that subjects will not be excluded from enrollment onto this study if their urine test is positive for drugs on initial screening. The following guidelines will be followed for positive drug screens on study procedure days:

      * If a Healthy Volunteer subject s urine drug screen test is positive on days involving imaging (MRI and/or PET) and NP testing, the procedures will be postponed and rescheduled. We will allow for up to 3 rescheduled study days resulting from positive urine drug screens. If the drug test is positive on the third rescheduled visit, the participant will be withdrawn from the study.
      * If a CUD subject s urine drug screen test is positive for drugs (except cocaine), the procedures will be postponed and rescheduled to another day. We will not place a limit on rescheduling study days in this participant group.

        * Note: At any time a subject expresses that he/she wants to get treatment for their cocaine use, we will immediately refer him/her to a treatment program. The subject will be withdrawn from the study at that time.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
To determine if there is disruption in circadian rhythms in cocaine use disorder (CUD) as compared to healthy controls. | end of study
  To assess if there are diurnal rhythms in DA signaling and in reward brain circuits and to determine if these are disrupted in cocaine addiction.

SECONDARY OUTCOMES:
Measuring dopamine signaling | end of study
  To assess if DA signaling correlates with reactivity of brain reward regions to exposure of drug and with functional connectivity of thereward network and to assess if the reactivity of reward network shows circadian variability.
Measuring circadian typology | end of study
  To determine if differences in the measures of DA signaling between morning and evening correlate with circadian typology.
Measuring sleep patterns | end of study
  To determine if measures of DA signaling correlate with measures of spontaneous motor activity and with sleeping patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Gene-Jack Wang, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.Data is analyzed by subject group and not on an individual basis.

REFERENCES:
- [Background] Wang GJ, Volkow ND, Fowler JS, Logan J, Pappas NR, Wong CT, Hitzemann RJ, Netusil N. Reproducibility of repeated measures of endogenous dopamine competition with [11C]raclopride in the human brain in response to methylphenidate. J Nucl Med. 1999 Aug;40(8):1285-91. PMID 10450679
- [Background] Wang GJ, Volkow ND, Logan J, Pappas NR, Wong CT, Zhu W, Netusil N, Fowler JS. Brain dopamine and obesity. Lancet. 2001 Feb 3;357(9253):354-7. doi: 10.1016/s0140-6736(00)03643-6. PMID 11210998
- [Background] Dunn JP, Cowan RL, Volkow ND, Feurer ID, Li R, Williams DB, Kessler RM, Abumrad NN. Decreased dopamine type 2 receptor availability after bariatric surgery: preliminary findings. Brain Res. 2010 Sep 2;1350:123-30. doi: 10.1016/j.brainres.2010.03.064. Epub 2010 Mar 31. PMID 20362560
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-AA-0187.html